CLINICAL TRIAL: NCT05406245
Title: The Effect of Stress on the Residual Gastric Volume in Older Adults Undergoing Staged-bilateral Total Knee Arthroplasty After Drinking Carbohydrate-containing Fluids: A Prospective Observational Study
Brief Title: The Effect of Stress on the Residual Gastric Volume
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Hyo-Seok Na, Professor, Seoul National University Bundang Hospital
Other Study IDs: B-2206-761-301
Record Dates: First submitted 2022-06-01; First posted 2022-06-06 (Actual); Last update posted 2022-07-05 (Actual); Status verified 2022-07

CONDITIONS: Arthritis Knee

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group C: Patients drank carbohydrate fluid 2 hours prior to surgery.
  Interventions: Dietary Supplement: Carbohydrate drinking

INTERVENTIONS:
Dietary Supplement: Carbohydrate drinking — Administration of carbohydrate fluid

SUMMARY:
In our institution, many patients undergo staged bilateral total knee arthroplasty at weekly intervals, and most of the patients are older adults with degenerative arthritis. As recommended, the older adult patients who undergoing total knee arthroplasty drink carbohydrate-containing fluid (400 ml) 2 hours prior to surgery. In this type of surgery, there are additional points to consider when applying the fasting guidelines. This is because, in addition to the factor of advanced age, which can affect gastric emptying time, the patient's physical, medical, and psychological conditions at the first and the second operation may be different. For example, the effect of the acute pain that occurs after the first total knee arthroplasty and subsequent opioids administered on gastric motility cannot be ignored. However, to date, there have been no studies examining the association of stress (emotional and surgical) and residual gastric volume of older adult patients with staged bilateral total knee arthroplasty and whether there is a difference according to the stage when carbohydrate-containing fluid is ingested.

In the present study, the investigators will evaluate the effect of emotional stress, surgical stress, pain, and the use of opioids on the residual gastric volume in older adults undergoing staged-bilateral total knee arthroplasty.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for staged bilateral total knee arthroplasty aged ≥ 65
* American Society of Anesthesiologists physical status classification 1, 2, and 3
* Body mass index < 35 kg/cm2
* Patients administered carbohydrate-containing fluid 2 hours prior to surgery

Exclusion Criteria:

* Previous surgery of the upper gastrointestinal tract
* Achalasia
* Diabetes

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Study participants will be patients who are scheduled to undergo staged bilateral total knee arthroplasty requiring administration of carbohydrate-containing fluid 2 hours prior to surgery.
Sampling Method: Non-Probability Sample
Enrollment: 53 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2023-09-15 (Estimated); Study Completion 2023-12-15 (Estimated)

PRIMARY OUTCOMES:
Level of stress hormone 1 | After induction of spinal anesthesia at first stage total knee arthroplasty/ an average 10 minutes
  Stress hormone (interleukin-1β, interleukin-6, interleukin-10, and tumor necrosis factor-α) measured after induction of spinal anesthesia
Level of stress hormone 2 | After induction of spinal anesthesia at second stage total knee arthroplasty/ an average 10 minutes
  Stress hormone (interleukin-1β, interleukin-6, interleukin-10, and tumor necrosis factor-α) measured after induction of spinal anesthesia

SECONDARY OUTCOMES:
Gastric volume 1 | First stage operation, during the gastric volume measuring at preoperative holding area/ an average of 30 minutes
  Gastric volume measured before induction of spinal anesthesia using ultrasound
Gastric volume 2 | Second stage operation, during the gastric volume measuring at preoperative holding area/ an average of 30 minutes
  Gastric volume measured before induction of spinal anesthesia using ultrasound
Anxiety scale 1 | First stage operation, one day before surgery/ an average of 30 minutes
  Anxiety scale measured before surgery
Anxiety scale 2 | Second stage operation, one day before surgery/ an average of 30 minutes
  Anxiety scale measured before surgery

CONTACTS AND LOCATIONS:
Overall Officials: Hyo-Seok Na, MD., PhD., Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No